CLINICAL TRIAL: NCT07184112
Title: Bridging the Gap Between Theory and Practice: Evaluating Embedded Micro-Scenarios in Simulation on Academic Motivation and Clinical Decision-Making Among Nursing Students-A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Assistant Professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HPO-05-FT-25/16
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Clinical Decision-Making in Nursing; Academic Motivation Scale
Keywords: Academic Motivation; Clinical Decision-Making; Nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micro-Scenarios (Experimental): The Embedded Micro-Scenario Simulations (EMSS) for nursing students include a series of engaging clinical cases designed to bridge the theory-practice gap.
  Interventions: Behavioral: The Embedded Micro-Scenario Simulations (EMSS)
- Control (Active Comparator): Routine teaching
  Interventions: Behavioral: The Embedded Micro-Scenario Simulations (EMSS)

INTERVENTIONS:
Behavioral: The Embedded Micro-Scenario Simulations (EMSS) — he Embedded Micro-Scenario Simulations (EMSS) for nursing students include a series of engaging clinical cases designed to bridge the theory-practice gap. In Prioritization of Care, students must prioritize three patients with varying degrees of urgency, honing their critical thinking skills. The Patient Education on Discharge scenario tasks them with effectively communicating self-care instructions. In End-of-Life Care, students provide compassionate support to a terminally ill patient and facilitate family discussions.

SUMMARY:
This study will utilize a convergent mixed-methods design. A quasi-experimental approach will be used to evaluate the effectiveness of EMSS in improving clinical decision-making skills among nursing students.

DETAILED DESCRIPTION:
This study will utilize a convergent mixed-methods design. A quasi-experimental approach will be used to evaluate the effectiveness of EMSS in improving clinical decision-making skills among nursing students.

The study will be conducted at the University of Hafr Albatin (UHB), located in Saudi Arabia. The institution is equipped with simulation labs and a digital learning management system, including access to a simulated EHR environment suitable for micro-scenario deployment.

ELIGIBILITY:
Inclusion Criteria:

Male undergraduate nursing students. Participants must possess basic computer literacy to effectively engage with the digital learning platform utilized in the simulation.

Exclusion Criteria:

* Female. non Saudi nursing students, students with mental health isssues

Ages: 18 Years to 27 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Decision-Making | 3 months
  This scale was originally developed by Jenkins (1983). Designed specifically for nursing students in the United States, the scale evaluates students' perceptions of clinical decision-making based on their self-reported experiences.
Academic Motivation | 3 months
  The Academic Motivation Scale (AMS) is the most popular tool for evaluating academic motivation. (Orsini et al., 2015). A 7-point Likert scale is used to rate each of the 28 items. The self-determination theory, which emphasizes the approach to human motivation and personality, is the theoretical foundation of the AMS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hafr Albatin, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No